CLINICAL TRIAL: NCT03483792
Title: Heritability of Polycystic Ovary Syndrome: Role of Antimullerian Hormone, Steroids and Leptin
Acronym: HERITOPK
Status: Completed | Type: Observational
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Other Study IDs: 2017_11; 2017-A02628-45 (Other: ID-RCB number, ANSM)
Record Dates: First submitted 2018-02-14; First posted 2018-03-30 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Polycystic Ovary Syndrome
Keywords: PCOS; AMH; Pregnancy; Heritability; LH
MeSH Terms: conditions — Polycystic Ovary Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — plasma placenta fragment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- PCOS group
  Interventions: Biological: Plasma dosage; Genetic: placental biopsy
- Control group
  Interventions: Biological: Plasma dosage; Genetic: placental biopsy

INTERVENTIONS:
Biological: Plasma dosage — 4 x 7 ml of blood punction at each control visit of the three trimesters of pregnancy
Genetic: placental biopsy — Immediately following delivery (<12h postpartum), placental biopsies (Collection of 4 placental fragments)

SUMMARY:
Polycystic ovary syndrome (PCOS) is the most common cause of ovulation disorders and affects 10 to 15% of women. Despite its frequency, its physiopathology remains unknown.

In women, Anti-Müllerian hormone (AMH) is secreted by granulosa cells located in the ovaries within the follicles. Compared to control women, serum AMH level is higher in PCOS women and could play a role in its pathophysiology. The severity of the PCOS phenotype is correlated with the production of AMH.

It is currently described in the literature that daughters of women with PCOS have a 50% risk of developing PCOS, but no genetic cause of transmission is known. In mice (article in press), pregnant females injected with AMH give birth to offspring with PCOS symptoms. The AMH could thus also play a role in the heritability of PCOS in women. Our team demonstrated that AMH, in its active cleaved form, had a direct central action on the hypothalamus by increasing the pulsatility of GnRH, inducing LH hypersecretion. The hypothesis is that AMH remains higher in pregnant women with PCOS and may affect the fetus by altering fetal and maternal hypothalamic secretions or by modifying placental steroid production.

Leptin has a role in reproduction, through its receptors located at the central (hypothalamus) and peripheral (granulosa cells) levels. In excessively high serum concentration, as observed in obesity, it would lead to a dysregulation of GnRH secretion, an alteration of ovarian steroidogenesis and a dysregulation of folliculogenesis.

Will be compare leptin levels in first trimester patients with and without PCOS to look for possible correlations between AMH and leptin and eliminate possible bias.

ELIGIBILITY:
Inclusion Criteria:

* Having a pre-conceptional infertility assessment in the gynecology-Endocrinology department of University Hospital of Lille
* in the first trimester of mono fetal pregnancy (between 5 and 10 weeks of gestation), obtained spontaneously, after induction of ovulation or Assisted Reproductive Techniques (ART)
* Pregnancy followed at University Hospital of Lille
* PCOS group: defined according to modified Rotterdam criteria (2003 and 2011)
* At least 2 of the following 3 criterion:

  * Cycle disorder
  * Clinical and / or biological hyperandrogenism
  * Ovarian volume > 10cm³ and/or more than 19 follicles from 2 to 9 mm per ovary
* After exclusion of other causes of cycle disorder or hyperandrogenism
* Control group: patient with severe male and / or tubal infertility, no cycling disorder, normal ovarian reserve (FSH<10 IU / L, E2<50 pg / ml, AMH>7 and <35 pmol / L and Follicles count between >5 and <20 per ovary at day 3 of the cycle).

In the group of female controls, the fertility problem is not related to a female pathology of the hypothalamic-pituitary-ovarian axis (tubal or male infertility). They are women without ovarian personal pathology. The problem of fertility being of other origin.

Exclusion Criteria:

* Multiple pregnancy
* Pregnancy after egg donation
* Long-term drug therapy (excluding routine pregnancy supplementation)
* Previous Diabetes
* Bariatric surgery
* Patients with ovulatory infertility of central or idiopathic origin
* Patients already included in another protocol

Ages: 18 Years to 43 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Study Population: Patients having a pre-conceptionnal infertility assessment in the gynecology-Endocrinology department of the CHRU of Lille, in the first trimester of monofetal pregnancy (between 5 and 10 weeks of gestation), obtained spontaneously, after induction of ovulation or Assisted Reproductive Techniques (ART)
Sampling Method: Non-Probability Sample
Enrollment: 58 (Actual)
Dates: Start 2018-04-20 (Actual); Primary Completion 2022-06-02 (Actual); Study Completion 2022-06-02 (Actual)

PRIMARY OUTCOMES:
Rate of plasma AMH in the 3rd trimester of pregnancy | between 29 and 44 amenorrhea weeks

SECONDARY OUTCOMES:
The variation of maternal plasma AMH | At baseline, between 5 and 15 amenorrhea weeks, between 15+1 day and 28+ 6 days amenorrhea weeks, between 29 and 44 amenorrhea weeks
The percentage change in the different forms of AMH (pro-AMH and cleaved forms) | At baseline, between 5 and 15 amenorrhea weeks, between 15+1 day and 28+ 6 days amenorrhea weeks, between 29 and 44 amenorrhea weeks
The variation in oestradiol, testosterone and LH levels | At baseline, between 5 and 15 amenorrhea weeks, between 15+1 day and 28+ 6 days amenorrhea weeks, between 29 and 44 amenorrhea weeks
The rate of leptin (only dosage in fasting patients) | between 5 and 15 amenorrhea weeks
The level of expression of aromatase, AMH and AMH Receptor II in the placenta | at delivery

CONTACTS AND LOCATIONS:
Overall Officials: Sophie Catteau-Jonard, MD,PhD, Principal Investigator — University Hospital, Lille
Locations (1):
- Hôpital Jeanne de Flandres, CHU, Lille, France

REFERENCES:
- [Result] Peigne M, Simon V, Pigny P, Mimouni NEH, Martin C, Dewailly D, Catteau-Jonard S, Giacobini P. Changes in circulating forms of anti-Muullerian hormone and androgens in women with and without PCOS: a systematic longitudinal study throughout pregnancy. Hum Reprod. 2023 May 2;38(5):938-950. doi: 10.1093/humrep/dead050. PMID 36921289